CLINICAL TRIAL: NCT02965638
Title: A Pilot Randomized Controlled Trial of Maternal Oxygen Therapy for Fetal Left Heart Hypoplasia
Brief Title: Trial of Maternal Oxygen for Fetal Left Heart Hypoplasia
Acronym: P-RCT-MHO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaine Morris (Other)
Responsible Party: Sponsor-Investigator, Shaine Morris, Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H37471
Record Dates: First submitted 2016-11-10; First posted 2016-11-17 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Fetal Left Heart Hypoplasia
Keywords: LHH
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen Group (Active Comparator): The mothers will be asked to be on 4 liter of oxygen through nasal cannula up to 24 hours a day. The subjects will be blinded to their treatment.
  Interventions: Other: Oxygen
- Control Group (No Intervention): These mothers will not undergo CMH therapy

INTERVENTIONS:
Other: Oxygen — The intervention arm (Oxygen Group) will receive oxygen via nasal cannula at a rate of 4L of FiO2 93-100% from an oxygen concentrator up to 24 hours daily
  Arms: Oxygen Group

SUMMARY:
The purpose of this study is to determine if maternal hyperoxygenation is an effective treatment for fetal left heart hypoplasia versus room air (placebo). This will be determined by measuring how well a baby's heart valves and their surrounding tissue are growing and functioning.

In addition the investigators will examine brain growth using fetal ultrasound and MRI, and MRI of the child's brain after they are born to determine if there is greater neonatal brain maturity or mothers receiving oxygen compared to fetuses of mothers not receiving oxygen.

Of note, the trial was initially randomized. However, due to low sample size and hesitation about randomization, the trial was converted to an open label study, allowing families opting for oxygen therapy to be in the intervention arm.

DETAILED DESCRIPTION:
Birth defects are the leading cause of infant mortality in the United States, and congenital heart disease is the leading cause of birth-defect related infant mortality. Despite advances, conditions related to left heart hypoplasia (LHH) are the most severe, and contribute significantly to this overall mortality as well as morbidity, including delayed brain maturation.

Conditions involving left heart hypoplasia (LHH) are among the most severe, and contribute significantly to this overall mortality. Sequelae are not limited to mortality, as recurrent interventions and impaired neurodevelopmental outcomes are highly prevalent among survivors with LHH. During the last 15 years, fetal cardiac intervention (FCI) has been introduced as a novel treatment for these children. The potential to halt disease progression in utero and to avoid or reduce the complexity of future surgery is very alluring. Current FCI is highly invasive, and there is limited and controversial data pertaining to efficacy, risk, and criteria for intervention. There is also a group of fetuses with LHH who require neonatal intervention, which may include single ventricle palliation, but are not candidates for current FCI.

The investigators intend to use a pilot study design to evaluate a novel non-invasive FCI to improve left heart growth in the fetus with LHH. The intervention will be chronic administration of supplemental oxygen provided to pregnant subjects (maternal hyperoxygenation, MH) compared to subjects not undergoing MH. Currently, two FCIs are available for left-sided disease, both of which are invasive and carry significant risk. The interventions include aortic valvuloplasty for aortic stenosis and atrial septoplasty/stenting for hypoplastic left heart syndrome with a restrictive or intact atrial septum. While there is tremendous enthusiasm for these procedures, there is limited and controversial data pertaining to efficacy, risk, and inclusion criteria for intervention.

There is also a further group of patients with LHH without frank aortic stenosis but hypoplasia of multiple left heart structures. While these patients almost universally require neonatal intervention which may include single ventricle palliation, they are not candidates for the fetal interventions currently available. This is the population of fetuses that we intend to target. The etiologies of left heart obstruction are unknown, although the common pathway is thought to be diminished blood flow to left heart structures in utero. Hypothesized etiologies include abnormal or restricted PFO flow, reduced flow across the mitral valve atrial septal aneurysm, low aortic flow due to aortic valvar abnormalities, presence of a ventricular septal defect, or subaortic narrowing. In the fetus, maternal blood with the highest oxygen and glucose concentration is delivered via the umbilical, and travels via the ductus venosus to the right atrium, where the majority crosses the foramen ovale and passes to the left heart. Most of that blood is used to perfuse the developing brain. In the normal fetal heart, about 10% of the left heart output, rather than traveling to the cerebral circulation, passes through the aortic isthmus and joins the blood that will perfuse the lower body. The low volume of blood flow through the fetal lungs is due to high pulmonary vascular resistance. The fetal pulmonary circulation is very sensitive to small changes in pulmonary arterial oxygen saturation and tension. Pulmonary vascular responses to changes in oxygen levels are very much related to gestational age and this sensitivity increases dramatically with advancing gestational age in the fetus.

It has been shown in both fetal sheep and human fetuses that when supplemental oxygen is provided to gravid mothers, there is evidence of an increase in fetal pulmonary blood flow, and this response becomes more pronounced late in gestation. This increase in pulmonary blood flow results in greater blood flow to the left atrium, and potentially to the left ventricle and across the aorta.

From January 2013 to March 2014 , the investigators conducted a pilot feasibility study of CMH in mothers of fetuses with LHH defined as a combined aortic & mitral valve annuli z-score (AMZ) less than -4.5. The investigators recruited gravidae with moderate to severe hypoplasia of left heart structures in which growth potential still existed; therefore gravidae with fetal hypoplastic left heart syndrome or severe aortic stenosis were excluded. Candidates were challenged as follows: After a full fetal echocardiogram in room air, Doppler scans were repeated after 10 minutes of maternal hyperoxygenation at 8 LPM 100% FiO2. Responders (fetuses with greater than 10% increase in aortic/combined cardiac output) were offered enrollment. Nine gravidae were enrolled. Chronic MH consisted of a minimum of 8 hours daily oxygen until delivery. Enrolled gravidae were compared to retrospective controls, who were all cared for at our institution from January 2013 to March 2014 with fetal LHH not undergoing CMH (9 total). Rate of growth in aortic and mitral annuli was compared among groups using longitudinal regression.

All mothers tolerated CMH, and there were no significant maternal or fetal complications. Mean increase in percent aortic flow after acute maternal hyperoxygenation was 35.3% (range 18.1-47.9%). Mean daily CMH hours = 10 (range 6.5-14.6). Mitral annular growth was 0.19 mm/week compared to 0.14 mm/week in CMH vs. controls (p=0.33). Aortic annular growth was 0.14 mm/week compared to 0.13 mm/week in CMH vs. controls (p=0.75). More than 9 CMH hours daily was associated with better growth of the aortic annulus in intervention fetuses (0.16 mm/week vs. 0.08 mm/week, p=0.014). In this pilot study, CMH appears safe and feasible, although effect estimates of annular growth were small given the studied method of delivery and dose of oxygen.

Given these findings, the investigators determined that CMH therapy should be further investigated as a low risk intervention for fetal LHH. The current study design is a pilot open label trial, with a change in the route and dose of oxygen as illustrated below.

Purpose and Objectives The investigators aim to perform a pilot trial to investigate the novel fetal cardiac intervention of continuous supplemental oxygen (maternal hyperoxygenation or MH) to mothers of fetuses with left heart hypoplasia (LHH). It has been shown that with acute MH, there is evidence of an increase in fetal pulmonary blood flow resulting in greater blood flow to the left atrium, left ventricle and across the aorta. There is evidence that chronic MH (CMH) in fetuses with hypoplastic left heart structures may improve growth of the left heart, although these studies did not include control patients. CMH also has the potential to attenuate prenatal cerebral changes thought to be secondary abnormal cerebral blood delivery in fetuses with LHH and resultant poor maturation of the fetal brain.

For the pilot study, the investigators intend to compare CMH to those without CMH in 12 mothers to determine effect estimates for a larger, multicenter randomized control trial (RCT) trial. The team has completed a feasibility pilot in which 9 mothers received CMH therapy. While there were no significant maternal or fetal complications, and results were promising, effect estimates were small and controls were only retrospective, and not randomized, limiting the interpretability of effect.

Aim 1: To determine if CMH therapy in mothers of fetuses with left heart hypoplasia results in faster growth of the fetal mitral and aortic annuli compared to fetuses of mothers with no CMH therapy. Methods & approach: Recruitment will include mothers of fetuses with LHH. Enrollees will wear a nasal cannula with 4 LPM flow 40% FiO2 oxygen or room air for 24 hours/day. Fetuses will be followed with echocardiography until delivery, when they will have an echocardiogram at birth, and further care as clinically indicated. Rates of change in left-sided valve annular dimensions in the CMH group vs. the non-CMH will be compared, using longitudinal regression.

Aim 2: To determine if CMH therapy in mothers of fetuses with left heart hypoplasia results in greater neonatal brain maturity compared to fetuses of mothers receiving no CMH. Methods & approach: Recruitment, enrollment, and the intervention are identical to that delineated above, as these will be the same patients. For this aim, brain maturity in fetuses exposed to MH versus no CMH will be compared using neonatal brain magnetic resonance imaging, as defined by a well-known maturation score.

CMH for fetal LHH has the potential to have a major impact in the field of congenital heart disease, as it is noninvasive, inexpensive, and universally available. Other institutions in the United States and Canada have demonstrated eagerness to join in a multicenter RCT if the pilot suggests positive results.

ELIGIBILITY:
Inclusion Criteria:

Mothers carrying fetuses with small left sided structures likely needing neonatal intervention, defined as the following on fetal echocardiography:

1. Sum of aortic and mitral valve z-scores (standard deviation based on gestational age) less than -4.5
2. Flow across the atrial septum either bidirectional or left to right
3. Transverse aortic arch or isthmus z-score less than 2.0.

Exclusion Criteria:

1. Severe fetal aortic stenosis
2. Fetal mitral or aortic atresia
3. Abnormal fetal atrioventricular or ventriculoarterial relationships, including double inlet left ventricle, double outlet right ventricle, transposition of the great arteries
4. Multiple gestations
5. Intrauterine growth restriction
6. Persistent fetal arrhythmia
7. Very poor ultrasound images, defined by the inability to reliably measure/evaluate all included cardiac structures
8. Major fetal extracardiac anomalies, specifically lesions that would be expected toi ncrease mortality for the fetus/neonate or would necessitate intervention in the neonatal period, including but not limited to congenital diaphragmatic hernia, omphalocele, gastroschesis, meningomyelocele, lower urinary tract obstruction, and anencephaly
9. Aneuploidy (although this is not required to be known to enroll
10. Maternal conditions that may alter fetal hemodynamic, including moderate to severe hypertension requiring medication in pregnancy, preeclampsia, major or unrepaired maternal congenital heart disease, obstructive sleep apnea, severe asthma (requiring daily treatment), restrictive lung disease, severe anemia (hemoglobin less than 8 g/dL), maternal chronic renal disease (creatinine greater than 1.2 mg/dL), known placental abnormality (complete placenta previa, accrete, or percreta), and antiphospholipid antibody syndrome.

Ages: 14 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-09; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Fetal aortic valve growth | from study enrollment to delivery
  The rate of growth of the fetal aortic valve using fetal echocardiography during serial echocardiography throughout enrollment during the fetal period
Fetal mitral valve growth | from study enrollment to delivery
  The rate of growth of the fetal mitral valve using fetal echocardiography during serial echocardiography throughout enrollment during the fetal period

SECONDARY OUTCOMES:
Brain maturation score by cerebral magnetic resonance imaging | performed after birth prior to cardiac surgery if necessary, which will be within the first 30 days of life
  Measured from postnatal Brain MRI
Neurologic injury on postnatal brain MRI | performed after birth prior to cardiac surgery if necessary, which will be within the first 30 days of life
  Evaluated on postnatal Brain MRI
Neurodevelopmental assessments | at 6 and 12 months
  Series of neurodevelopmental tests
Change in measured parameters on fetal neurosonography and fetal brain MRI | from study enrollment to delivery
  neurosonography during serial examinations throughout enrollment during the fetal period

CONTACTS AND LOCATIONS:
Overall Officials: Shaine A Morris, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No.

REFERENCES:
- [Background] Lara DA, Morris SA, Maskatia SA, Challman M, Nguyen M, Feagin DK, Schoppe L, Zhang J, Bhatt A, Sexson-Tejtel SK, Lopez KN, Lawrence EJ, Andreas S, Wang Y, Belfort MA, Ruano R, Ayres NA, Altman CA, Aagaard KM, Becker J. Pilot study of chronic maternal hyperoxygenation and effect on aortic and mitral valve annular dimensions in fetuses with left heart hypoplasia. Ultrasound Obstet Gynecol. 2016 Sep;48(3):365-72. doi: 10.1002/uog.15846. PMID 26700848